CLINICAL TRIAL: NCT03580863
Title: Coverage and Future of Children Referred by a Liberal Doctor's Letter to Pediatric Emergency in Strasbourg Teaching Hospital Compared With Children Who Are Coming by Themselves in 2017
Brief Title: Referred vs Spontaneous Visits at Pediatric ER: an Outcome Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7008
Record Dates: First submitted 2018-06-14; First posted 2018-07-09 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-01

CONDITIONS: Emergency Surgical
Keywords: Pediatric; emergency surgical and medical service; Liberal doctor; complaint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since 80's, admissions in Emergency medical services increase regularly. Children represents 30% of the patients in Emergency medical Service. Only 20% of admissions are hospitalized and only 3 % need emergency care. Consequences are team's exhaustion, a reduction of healthcare quality, a slowdown in emergency care.

Investigator decided to realize an epidemiologic prospective study in Emergency medical and surgical Pediatric Service in Strasbourg Teaching Hospital to compare coverage of children who are referred by a liberal doctor with children who are coming by themselves matched with age and complaint.

This study will analyze the relevance of complaints and decision-making factors for the liberal doctor to send children in Emergency Medical and Surgical Service. Investigator will talk about the importance of close collaboration between liberal doctor and hospital doctor, as well as patient's information about basic care service on nights and week-ends in order to decrease the number of emergency admission.

ELIGIBILITY:
Inclusion Criteria:

* Any child attending the pediatric medical and surgical emergency department of Strasbourg University Hospital, accompanied by at least one of his parents.
* Age of the patient: from birth to 18 years.
* Patient sent by mail from a liberal doctor (general practitioner, liberal pediatrician, PMI, SOS doctor ...) for the first group.
* Or emergency consultant spontaneously for the second group.
* Understanding and speaking French
* Having agreed to participate in the study if it is old, or whose parents have agreed to participate in the study.

Exclusion Criteria:

* Patient unaccompanied by one of his parents
* Refusal to participate in the study.
* Vital emergency or immediate care needed
* Patient arriving at the emergency department at first alone with paramedics or the SMUR, then joined by his parents secondarily
* Patients referred by a liberal doctor but without mail.

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: * Any child attending the pediatric medical and surgical emergency department of Strasbourg University Hospital, accompanied by at least one of his parents.
  * Age of the patient: from birth to 18 years.
  * Patient sent by mail from a liberal doctor (general practitioner, liberal pediatrician, PMI, SOS doctor ...) for the first group.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of hospitalization frequency | The period from January 1st, 2016 to December 31st, 2017 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Dimitar TCHOMAKOV, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service D'Urgences Medico Chirurgicales Pediatriques, Strasbourg, France